CLINICAL TRIAL: NCT04699188
Title: A Phase Ib/II Open-label, Multi-center Dose Escalation Study of JDQ443 in Patients With Advanced Solid Tumors Harboring the KRAS G12C Mutation
Brief Title: Study of JDQ443 in Patients With Advanced Solid Tumors Harboring the KRAS G12C Mutation
Acronym: KontRASt-01
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CJDQ443A12101; 2020-004129-22 (EudraCT Number)
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: KRAS G12C Mutant Solid Tumors; Carcinoma, Non-Small-Cell Lung; Carcinoma, Colorectal; Cancer of Lung; Cancer of the Lung; Lung Cancer; Neoplasms, Lung; Neoplasms, Pulmonary; Pulmonary Cancer; Pulmonary Neoplasms
Keywords: KRAS; KRAS G12C; Metastatic cancer; Advanced cancer; Enzyme inhibitor; PD-1; SHP2; Targeted therapy; Non-small-cell lung cancer; colorectal cancer; Molecular mechanisms of pharmacological action
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Lung Neoplasms; Neoplasm Metastasis | interventions — JDQ443; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (Experimental): JDQ443
  Interventions: Drug: JDQ443
- Arm B (Experimental): JDQ443 in combination with TNO155
  Interventions: Drug: JDQ443; Drug: TNO155
- Arm C (Experimental): JDQ443 in combination with tislelizumab
  Interventions: Drug: JDQ443; Biological: tislelizumab
- Arm D (Experimental): JDQ443 in combination with TNO155 and tislelizumab
  Interventions: Drug: JDQ443; Drug: TNO155; Biological: tislelizumab

INTERVENTIONS:
Drug: JDQ443 — KRAS G12C inhibitor
Drug: TNO155 — SHP2 inhibitor
  Arms: Arm B; Arm D
Biological: tislelizumab — Anti PD1 antibody
  Arms: Arm C; Arm D

SUMMARY:
This is a phase Ib/II open label study. The escalation part will characterize the safety and tolerability of JDQ443 single agent and JDQ443 in combination with the other study treatments (TNO155 and tislelizumab) in advanced solid tumor patients. After the determination of the maximum tolerated dose / recommended dose for a particular treatment arm, dose expansion will assess the anti-tumor activity and further assess the safety, tolerability, and PK/PD of each regimen at the maximum tolerated dose / recommended dose or lower dose.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with advanced (metastatic or unresectable) KRAS G12C mutant solid tumors who have received standard of care or are intolerant or ineligible to approved therapies
* ECOG Performance Status of 0 or 1
* At least one measurable lesion as defined by RECIST 1.1
* Prior treatment with a KRAS G12C inhibitor may be allowed for dose escalations of combinations and a subset of groups in dose expansion

Exclusion Criteria:

* Tumors harboring driver mutations that have approved targeted therapies, with the exception of KRAS G12C mutations
* Symptomatic brain metastases or known leptomeningeal disease. Patients with asymptomatic treated or untreated brain metastases may be eligible
* Clinically significant cardiac disease or risk factors at screening
* A medical condition that results in increased photosensitivity Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2026-08-26 (Estimated); Study Completion 2026-08-26 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Incidence and severity of dose limiting toxicities (DLTs) during the first cycle of monotherapy or combination treatment | 21 days
  A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first cycle of treatment
Dose Escalation: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | 24 months
  All information obtained on AE will be displayed by treatment group. Summary tables will include only AEs that started/worsened during the cycles of treatment (treatment-emergent AEs).
Dose Escalation: Frequency of dose interruptions and reductions, by treatment | 24 months
  Tolerability of study drug will be assessed by summarizing the number of and reason for dose delays and dose reductions.
Dose Escalation: Dose intensity by treatment | 24 months
  Dose intensity is defined as the ratio of actual cumulative dose received and actual duration of treatment.
Dose Expansion: Overall response rate (ORR) per RECIST v1.1, by treatment | 24 months
  Overall response rate is defined as the proportion of patients with a BOR of CR or PR according to RECIST 1.1, and will be summarized along with the corresponding 95% exact binomial confidence interval (CI). Applies to all groups except the brain metastasis group.
Dose expansion: Overall intracranial response rate (OIRR) per mRANO-BM | 24 months
  OIRR per mRANO-BM is defined as the proportion of participants with a best overall intracranial response (BOIR) of CR or PR according to mRANO-BM criteria, and will be summarized along with the corresponding 90% and 95% exact CI. Applies to brain metastasis group only.
Dose expansion: Incidence and severity of AEs and SAEs | 24 months
  All information obtained on AE will be displayed by treatment group. Summary tables will include only AEs that started/worsened during the cycles of treatment (treatment-emergent AEs). Applies to JDQ443 dose randomization group only.
Dose expansion: frequency of dose interruptions and reductions, by treatment | 24 months
  Tolerability of study drug will be assessed by summarizing the number of and reason for dose delays and dose reductions. Applies to JDQ443 dose randomization group only.
Dose expansion: Dose intensity by treatment | 24 months
  Dose intensity is defined as the ratio of actual cumulative dose received and actual duration of treatment. Applies to JDQ443 dose randomization group only
Dose expansion: ORR per RECIST 1.1 of JDQ443 single agent in patients with non-small cell lung cancer (JDQ443 dose randomization group only) | 24 months
  Overall response rate is defined as the proportion of patients with BOR of CR or PR according to RECIST 1.1, and will be summarized along with the corresponding 95% exact binomial confidence interval (CI). Applies to JDQ443 dose randomization group only

SECONDARY OUTCOMES:
Dose Escalation and Expansion: ORR per RECIST v1.1 | 24 months
  Overall response rate is defined as the proportion of patients with a BOR of CR or PR according to RECIST 1.1, and will be summarized along with the corresponding 95% exact binomial confidence interval (CI)
Dose Escalation and Expansion: Best Overall Response (BOR) per RECIST v1.1 | 24 months
  BOR is defined as the best overall confirmed response recorded from the start of the treatment until disease progression/recurrence.
Dose Escalation and Expansion: Progression-free survival (PFS) per RECIST v1.1, Overall Survival (OS) | 24 months
  Per RECIST 1.1, PFS is defined as the time from the date of start of treatment to the date of the first documented progression, or death. If patient has not had an event, PFS will be censored at the date of last adequate tumor assessment. PFS will be summarized using the Kaplan-Meier method, along with 95% CI
Dose Escalation and Expansion: Duration of Response (DOR) per RECIST v1.1 | 24 months
  Duration of response is defined as the time from the date of the first documented response (CR or PR), to the date of first documented progression, or death due any cause. Estimates will use Kaplan-Meier method, and median DOR and corresponding 95% CI will be presented.
Dose Escalation and Expansion: Disease Control Rate (DCR) per RECIST v1.1 | 24 months
  The disease control rate is calculated as the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease. It will be summarized along with the corresponding 95% exact CI
Dose Escalation and Expansion: Plasma or serum concentration vs time profiles (AUC) by treatment | Up to 24 months
  AUC is defined as area under the plasma or serum concentration versus time curve after a dose of JDQ443, TNO155 and tislelizumab
Dose Escalation and Expansion: Plasma concentration (Cmax) by treatment | Up to 24 months
  Cmax is defined as the maximum observed plasma or serum drug concentration after single dose administration.
Dose Escalation and Expansion: Time to achieve Cmax (Tmax) by treatment | Up to 24 months
  Tmax is defined as the time to reach maximum plasma or serum drug concentration after single dose administration.
Dose Escalation and Expansion: Antidrug antibody (ADA) incidence by treatment | Up to 24 months
  To evaluate the immunogenicity of tislelizumab when dosed in combination with JDQ443 and/or TNO155 - only applicable to Arms C and D
Dose Expansion: Dose intensity by treatment | 24 months
Dose Expansion: Frequency of dose interruptions and reductions, by treatment | 24 months
  Tolerability of study drug will be assessed by summarizing the number of and reason for dose delays and dose reductions.
Dose Expansion: Incidence and severity of dose limiting toxicities (DLTs) during the first cycle of monotherapy or combination treatment | 21 days
  A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first cycle of treatment
Dose Expansion: Incidence and severity of AEs and SAEs by treatment | 24 months
Dose expansion: Intracranial disease control rate (IDCR) per mRANO-BM | 24 months
  IDCR is the proportion of participants with a confirmed BOIR of CR or PR or SD (or non-CR/non-PD) per mRANO-BM criteria. It will be summarized along with the corresponding 90% and 95% CI. Applies to the brain metastasis group only.
Dose expansion: Best overall intracranial response (BOIR) per mRANO-BM | 24 months
  BOIR is defined as the best overall confirmed response recorded from the start of the treatment until disease progression/recurrence per mRANO-BM, or until patient comes off study, whichever comes first. BOIR will be summarized along with the corresponding 95% exact CI. Applies to the brain metastasis group only.
Dose expansion: Intracranial progression free survival (IPFS) per mRANO-BM | 24 months
  IPFS is defined as the time from the date of start of treatment to the date of the first documented progression per mRANO-BM, or death due to any cause. If a patient has not had an event, IPFS will be censored at the date of last adequate tumor assessment. IPFS will be summarized using the Kaplan-Meier method. Median IPFS and IPFS probability at pre specified time-points will be presented along with 95% CI. Applies to the brain metastasis group only.
Dose expansion: Duration of intracranial response (DOIR) per mRANO-BM | 24 months
  DOIR is defined as the time from the date of first documented intracranial response of either CR or PR to the date of the first documented intracranial progression as per mRANO-BM criteria as assessed by central review or date of death due to underlying cause of cancer. DOIR will be summarized using the KM method if data permit. Median DOIR, with corresponding 95% CI. KM estimates for DOIR proportions at specific time points, along with 95% CI will also be provided. Applies to the brain metastasis group only.

CONTACTS AND LOCATIONS:
Locations (35):
- United States (4):
  - Emory University School of Medicine-Winship Cancer Institute, Atlanta, Georgia
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Uni Of TX MD Anderson Cancer Cntr, Houston, Texas
- Novartis Investigative Site, Melbourne, Victoria, Australia
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Montreal, Quebec, Canada
- China (2):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Beijing
- Novartis Investigative Site, Copenhagen, Denmark
- France (3):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Villejuif
- Germany (4):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Freiburg im Breisgau
- Novartis Investigative Site, Hong Kong, Hong Kong
- Italy (2):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Milan, MI
- Japan (5):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Koto Ku, Tokyo
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Spain (6):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Lorthiois E, Gerspacher M, Beyer KS, Vaupel A, Leblanc C, Stringer R, Weiss A, Wilcken R, Guthy DA, Lingel A, Bomio-Confaglia C, Machauer R, Rigollier P, Ottl J, Arz D, Bernet P, Desjonqueres G, Dussauge S, Kazic-Legueux M, Lozac'h MA, Mura C, Sorge M, Todorov M, Warin N, Zink F, Voshol H, Zecri FJ, Sedrani RC, Ostermann N, Brachmann SM, Cotesta S. JDQ443, a Structurally Novel, Pyrazole-Based, Covalent Inhibitor of KRASG12C for the Treatment of Solid Tumors. J Med Chem. 2022 Dec 22;65(24):16173-16203. doi: 10.1021/acs.jmedchem.2c01438. Epub 2022 Nov 18. PMID 36399068